CLINICAL TRIAL: NCT07372716
Title: Active Cancer Patients Having Cancer Related Invasive Procedures or Surgery and Needing Perioperative Management of Anticoagulation Therapy (ACE-HIGH): A Prospective Management Cohort Study
Brief Title: Safety of Perioperative Anticoagulation Management in People With Active Cancer Undergoing Cancer-Related Surgery or Procedures (ACE-HIGH Study)
Acronym: ACE-HIGH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACE-HIGH 20250647-01T
Record Dates: First submitted 2026-01-08; First posted 2026-01-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Thrombosis; Cancer; Thrombosis, Deep Vein; Atrial Fibrillation (AF); Venous Thromboembolic Event; Bleeding
Keywords: thrombosis; Atrial fibrillation; Cancer; Anticoagulant Interruption; VTE; bleeding
MeSH Terms: conditions — Thrombosis; Neoplasms; Venous Thrombosis; Atrial Fibrillation; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study intervention (Other): The intervention consists of applying perioperative anticoagulation management strategies based on contemporary guidelines for non-cancer patients to a cancer population undergoing invasive procedures or surgery. This study is a pragmatic, guideline-informed interventional study. It does not involve testing a novel drug, biologic, or device, and therefore does not align with clinical trial phases (Phase I-IV).
  Interventions: Other: standardized perioperative anticoagulation management Guideline

INTERVENTIONS:
Other: standardized perioperative anticoagulation management Guideline — The intervention is implementing a standardized perioperative anticoagulation management strategy in patients with active cancer (and this strategy is consistent with guideline-directed care for patients with active cancer).

SUMMARY:
The purpose of this study is to help find how safe current practices are when managing blood thinners in people with cancer who are having surgery or medical procedures. Investigators will also measure how often bleeding or clotting problems happen in this setting. The goal is to use this information to improve future care and reduce these risks for patients. This study will determine whether contemporary practices can be safely applied to cancer patients, and also evaluate the blood thinner level left over in patient's body at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Prescribed a Direct Oral Anticoagulant (DOAC), warfarin (International Normalized Ratio (INR) target 2.0-3.0) or Low Molecular Weight Heparin (LMWH) (75-100% weight-based therapeutic dosing) for stroke prevention in Atrial Fibrillation (AF) or the treatment of Venous Thromboembolism (VTE). Eligible DOAC regimens include full-dose (therapeutic) DOAC regimens appropriate for age and renal function. Eligible DOAC regimens include:

  i. Apixaban 10 mg po BID (VTE) ii. Apixaban 5 mg po BID (AF or VTE) iii. Apixaban 2.5 mg po BID (AF) iv. Rivaroxaban 15 mg po BID (VTE) v. Rivaroxaban 20 mg po OD (AF or VTE) vi. Rivaroxaban 15 mg po OD (AF only) vii. Edoxaban 60 mg po OD (AF or VTE) viii. Edoxaban 30 mg po OD (AF or VTE) ix. Dabigatran 150 mg po BID (AF or VTE) x. Dabigatran 110 mg po BID (AF)
* Has active cancer, defined as:

  i. cancer diagnosed within 6 months ii. recurrent, regionally advanced, or metastatic cancer iii. cancer for which treatment had been administered within 6 months before enrolment iv. hematologic cancer that is not in remission v. Patients who are felt to likely have active cancer based on clinical/imaging characteristics but are awaiting tissue confirmation and are scheduled for a biopsy procedure are eligible for trial inclusion
* Is undergoing a planned cancer-related inpatient or outpatient invasive procedure or cancer surgery (to diagnose, treat or palliate cancer; at investigator's discretion)
* Interruption of anticoagulation therapy for the planned procedure is required.

Exclusion Criteria:

* Presence of any mechanical prosthetic heart valve
* Known pregnancy or breastfeeding
* Severe renal insufficiency (Creatinine Clearance (CrCl) < 30 mL/min or < 25 mL/min for Apixaban users)
* Condition that might impair adherence to the study protocol (e.g., cognitive impairment, geographic inaccessibility) as determined by the treating physician
* Allergy to heparin or a history of (Heparin Induced Thrombocytopenia (HIT)
* More than one surgery/procedure planned during the study period
* Previous study participation
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Major bleeding events | From enrollment to the end of study follow ups at 4 weeks"
  Major bleeding is defined according to International Society on Thrombosis and Haemostasis (ISTH) criteria as any of the following within 30 days post-surgery:
  Fatal bleeding; OR Symptomatic bleeding in a critical area or organ (e.g., intracranial, intraspinal, intraocular, retroperitoneal, pericardial, non-operated joint, or intramuscular with compartment syndrome); OR Extrasurgical site bleeding causing ≥20 g/L hemoglobin drop or requiring ≥2 units of blood transfusion within 24-48 hours; OR Surgical site bleeding requiring re-intervention or causing delayed mobilization, prolonged hospitalization, or deep wound infection; OR Unexpected/prolonged surgical site bleeding causing hemodynamic instability with ≥20 g/L hemoglobin drop or transfusion of ≥2 units within 24 hours.

SECONDARY OUTCOMES:
30-day combined risk of ATE (Arterial Thromboembolism ) /VTE (Venous Thromboembolism) | 30 days
  Includes arterial or venous thromboembolic events: stroke, TIA (Transient Ischemic Attack), systemic embolism, DVT (Deep Venous Thromboembolism), PE (Pulmonary Embolism), splanchnic vein thrombosis, or cerebral venous sinus thrombosis.
30-day risk of clinically relevant non-major bleeding (ISTH definition) | 30 days
  Bleeding that does not meet major criteria but requires medical intervention, unscheduled contact with a physician, interruption of anticoagulation, or causes discomfort impacting daily activities.
30-day risk of all-cause mortality | 30 days
  Death from any cause within 30 days post-surgery
Time to resumption of anticoagulation (therapeutic dosing) | hours from surgery to administration of therapeutic anticoagulant dose.
  Measured in hours from surgery to administration of therapeutic anticoagulant dose.
Pre-operative residual anticoagulant levels | Perioperative/Periprocedural
  Measured at Visit #3 prior to surgery using drug-specific assays.
Pre-operative thrombin generation assay (TGA) parameters | Perioperative/Periprocedural
  Lag Time (in minutes)
Pre-operative thrombin generation assay (TGA) parameters | Perioperative/Periprocedural
  Time to Peak (in minutes)
Pre-operative thrombin generation assay (TGA) parameters | Perioperative/Periprocedural
  Peak thrombin generation (peak; in nM)
Pre-operative thrombin generation assay (TGA) parameters | Perioperative/Periprocedural
  Endogenous thrombin potential (ETP; in nM/min)
Pre-operative thrombin generation assay (TGA) parameters | Perioperative/Periprocedural
  Mean velocity rate index (mVRI; in nM/min).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Shaw, MD, MSc, FRCPC, Principal Investigator — Ottawa Hospital Research Institute